CLINICAL TRIAL: NCT03721718
Title: Phase I/IIa, Open-label, Dose Ranging Study to Evaluate the Safety, Tolerability and Immunogenicity of GLS-5300, Administered ID Followed by CELLECTRA® 2000 (Electroporation, EP)
Brief Title: Evaluate the Safety, Tolerability and Immunogenicity Study of GLS-5300 in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GeneOne Life Science, Inc. (Industry)
Collaborators: Inovio Pharmaceuticals (Industry); International Vaccine Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MERS-002
Record Dates: First submitted 2018-09-11; First posted 2018-10-26 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Healthy
Keywords: MERS CoV; MERS-CoV; Middle East Respiratory Syndrome; MERS; DNA Vaccine
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GLS-5300 with ID Cellectra electroporation (Experimental): GLS-5300 at 0.3mg DNA/dose
  Interventions: Biological: GLS-5300; Device: Cellectra 2000 Electroporation
- GLS-5300 at 0.3mg DNA/dose with ID Cellectra electroporation (Experimental): GLS-5300 at 0.3mg DNA/dose
  Interventions: Biological: GLS-5300; Device: Cellectra 2000 Electroporation
- GLS-5300 at 0.6mg DNA/dose (3 dose regimen) (Experimental): GLS-5300 at 0.6mg DNA/dose with ID Cellectra electroporation
  Interventions: Biological: GLS-5300; Device: Cellectra 2000 Electroporation
- GLS-5300 at 0.6mg DNA/dose (2 dose regimen) (Experimental): GLS-5300 at 0.6mg DNA/dose with ID Cellectra electroporation
  Interventions: Biological: GLS-5300; Device: Cellectra 2000 Electroporation

INTERVENTIONS:
Biological: GLS-5300 — [Part A] GLS-5300 0.3 mg at 0, 4, and 12 weeks (N=5) [Part B] GLS-5300 0.3 mg at 0, 4, and 12 weeks (N=5) GLS-5300 0.6 mg at 0, 4, and 12 weeks (N=25) GLS-5300 0.6 mg at 0 and 8 weeks (N=25)
Device: Cellectra 2000 Electroporation — GLS-5300 administered ID followed by Cellectra 2000 Electroporation

SUMMARY:
The Middle East Respiratory Syndrome Coronavirus (MERS CoV), is a cause of severe and highly fatal lower respiratory tract infection, first identified in 2012. As of August 2018, there have been 2229 cases reported with a case fatality rate >35%. In 2015 an individual returning to South Korea served as the index case for an outbreak of 186 individuals, of who, >20% died. GLS-5300 is a DNA plasmid vaccine that expresses the MERS CoV spike (S) glycoprotein. This Phase I/IIa study will evaluate the safety, tolerability and immunogenicity of GLS-5300 administered intradermally (ID) followed by electroporation at 0.3 and 0.6 mg/dose assessing 2 and 3-dose regimens.

DETAILED DESCRIPTION:
GLS-5300 is a DNA plasmid vaccine that expresses the MERS CoV spike (S) glycoprotein.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19-70 years;
2. Able to provide consent to participate and having signed an Informed Consent Form (ICF);
3. Able and willing to comply with all study procedures;
4. Women of child-bearing potential agree to either remain sexually abstinent, use medically effective contraception (oral contraception, barrier methods, spermicide, etc.) or have a partner who is sterile during this trials , or have a partner who is medically unable to induce pregnancy.
5. Normal screening ECG or screening ECG with no clinically significant findings;
6. Screening laboratory must be within normal limits or have only Grade 0-1 findings;
7. No history of clinically significant immunosuppressive or autoimmune disease.
8. Not currently or within the previous 4 weeks taking immunosuppressive agents (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or prednisone at a dose less than or equal to 10 mg/day or steroid equivalent).

Exclusion Criteria:

1. Administration of an investigational compound either currently or within 90 days of first dose;
2. Previous receipt of an investigational product for the treatment or prevention of MERS-CoV or SARS-CoV except if subject is verified to have received placebo;
3. Previous infection with MERS-CoV;
4. Administration of any vaccine within 4 weeks of first dose;
5. Administration of any monoclonal or polyclonal antibody product within 4 weeks of the first dose
6. Administration of any blood product within 3 months of first dose;
7. Pregnancy or breast feeding or plans to become pregnant during the course of the study;
8. History of positive serologic test for HIV, hepatitis B surface antigen (HBsAg); or any potentially communicable infectious disease as determined by the Principal Investigator or Medical Monitor;
9. Positive serologic test for HIV, Hepatitis B surface antigen, or hepatitis C (exception: successful treatment with confirmation of sustained virologic response);
10. Baseline evidence of kidney disease as measured by creatinine greater than 1.5mg/dL (CKD Stage II or greater);
11. Baseline screening lab(s) with Grade 2 or higher abnormality;
12. Chronic liver disease or cirrhosis;
13. Immunosuppressive illness including hematologic malignancy, history of solid organ or bone marrow transplantation;
14. Current or anticipated concomitant immunosuppressive therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or prednisone at a dose greater than 10 mg/day or steroid equivalent);
15. Past (within 6 months), current or anticipated treatment with TNF-α inhibitors such as infliximab, adalimumab, etanercept, or other monoclonal antibody;
16. Prior major surgery or any radiation therapy within 4 weeks of group assignment;
17. Any pre-excitation syndromes, e.g., Wolff-Parkinson-White syndrome; history of PSVT syndrome, history of prolonged QT syndrome;
18. Presence of a cardiac pacemaker or automatic implantable cardioverter defibrillator (AICD);
19. Metal implants within 20 cm of the planned site(s) of injection;
20. Presence of keloid scar formation or hypertrophic scar as a clinically significant medical condition at the planned site(s) of injection.
21. Prisoner or subjects who are compulsorily detained (involuntary incarceration) for treatment of either a physical or psychiatric illness;
22. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements or assessment of immunologic endpoints;
23. Not willing to allow storage and future use of samples for MERS-CoV related research
24. Any illness or condition that in the opinion of the investigator may affect the safety of the subject or the evaluation of any study endpoint.
25. Presence of tattoos covering all possible injection sites.
26. Healthcare workers participating in the medical examination of patients infection with MER

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Day0 through up to 60 weeks
  Incidence of Adverse events by System organ class (SOC); preferred term (PT); severity and relationship to study treatment and schedule
Administration (injection) site reactions | Day0 through up to 60 weeks
  Administration (injection) site reactions described by frequency
Changes in safety laboratory parameters | Day0 through up to 60 weeks
  Number of participants with changes based on frequency in safety lab parameters in Complete Blood Count and Liver panel tests" or similar.
Administration (injection) site pain | Administration (injection) site pain
  Administration (injection) site pain as described by Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Cellular Immune Responses | Day0 through up to 60 weeks
  Antigen specific cellular immune responses to MERS-CoV as determined by Interferon-gamma (IFN-γ) ELISpot
Binding antibody titers | Day0 through up to 60 weeks
  Binding antibody titers against MERS-CoV for a 2 and 3 dose vaccination regimens
Neutralizing antibodies | Day0 through up to 60 weeks
  Titers of neutralizing antibodies against MERS-CoV

CONTACTS AND LOCATIONS:
Overall Officials: Joel Maslow, MD, PhD, MBA, Study Chair — GeneOne Life Science, Inc.
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided